CLINICAL TRIAL: NCT06015919
Title: Effect of Dash Diet and Acupuncture on Hypertention in Postmenopausal Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Collaborators: faculty of physical therapy (Unknown)
Responsible Party: Principal Investigator, Alaa Nabil Elsayed Mohamed, principal investigator, Cairo University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P.T.REC/012/003872
Record Dates: First submitted 2023-02-10; First posted 2023-08-29 (Actual); Last update posted 2023-08-29 (Actual); Status verified 2023-08

CONDITIONS: Postmenopausal Disorder
MeSH Terms: interventions — Dietary Approaches To Stop Hypertension; Acupuncture Therapy

STUDY DESIGN:
Intervention Model Description: dash diet and acupuncture on post menopausal hypertention
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- effect of dash diet and acupuncture on hypertention in post menopausal women (Experimental): * Group (A): It will include 15 post-menopausal women who will be treated by DASH diet and anti-hypertensive drugs.
  * Group (B): It will include 15 post-menopausal women who will be treated by acupuncture and anti-hypertensive drugs.
  * Group (C): It will include 15 post-menopausal women who will be treated by DASH diet, acupuncture and anti-hypertensive drugs.
  Interventions: Behavioral: dash diet; Device: Acupuncture

INTERVENTIONS:
Behavioral: dash diet — * Group (A): It will include 15 post-menopausal women who will be treated by DASH diet and anti-hypertensive drugs.
  * Group (B): It will include 15 post-menopausal women who will be treated by acupuncture and anti-hypertensive drugs.
  * Group (C): It will include 15 post-menopausal women who will be treated by DASH diet, acupuncture and anti-hypertensive drugs.
Device: Acupuncture — acupuncture

SUMMARY:
A study of effect of dash diet and acupuncture on hypertension in postmenopausal women

DETAILED DESCRIPTION:
45 of post menopausal women divided into three groups A,B,C

* Group (A): It will include 15 post-menopausal women who will be treated by DASH diet and anti-hypertensive drugs.
* Group (B): It will include 15 post-menopausal women who will be treated by acupuncture and anti-hypertensive drugs.
* Group (C): It will include 15 post-menopausal women who will be treated by DASH diet, acupuncture and anti-hypertensive drugs.

ELIGIBILITY:
Inclusion Criteria:

* Their body mass index will be ranged from 25 -29.9 kg/m2
* All patients will be medically stable when attending the study.
* The DASH eating plan of 1800 kcal per day will be used in the study.

Exclusion Criteria:

* Auditory and visual problems.
* Chronic renal failure.
* Myocardial infarction or arrythmias with heart failure.

Ages: 50 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — post menopausal hypertensive women
Enrollment: 45 (Actual)
Dates: Start 2022-12-05 (Actual); Primary Completion 2023-04-25 (Actual); Study Completion 2023-08-20 (Actual)

PRIMARY OUTCOMES:
blood pressure | 3 months
  it will be measured by sphygmomanometer pre and post treatment

SECONDARY OUTCOMES:
sodium and potassium levels | 3 months
  it will be measured by blood analysis pre and post treatment

OTHER OUTCOMES:
assessment of quality of life | 3 months
  it will be measured by sf 36 questionnaire pre and post treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Alaa Nabil Elsayed Mohamed, Abū Ḩammād, Elsharqia, Egypt